CLINICAL TRIAL: NCT04183959
Title: Intubating Video Stylet Versus Fiberoptic Intubating Bronchoscope. A Randomised Comparative Study for Intubation in Lateral Position.
Brief Title: Intubating Video Stylet Versus Fiberoptic Intubating Bronchoscope.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Amr Samir Wahdan, Lecturer of Anesthesia, Pain management and Surgical ICU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MD-53-2019
Record Dates: First submitted 2019-11-29; First posted 2019-12-03 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Intubating Video Stylet
MeSH Terms: interventions — Optical Fibers

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group- video stylet intubation (VS) (Active Comparator): trachea will be intubated using laryngoscopic assisted video stylet device in lateral position
  Interventions: Device: video stylet
- Group- fiberoptic intubation (FO) (Active Comparator): : intubation will be done using fiberoptic device by the same anesthesiologist in lateral position
  Interventions: Device: fiberoptic

INTERVENTIONS:
Device: video stylet — trachea will be intubated using laryngoscopic assisted video stylet device in lateral position
  Arms: Group- video stylet intubation (VS)
Device: fiberoptic — intubation will be done using fiberoptic device by the same anesthesiologist in lateral position
  Arms: Group- fiberoptic intubation (FO)

SUMMARY:
the video stylet (VS), it is considered one of the newer devices in this category. It is a portable device with liquid crystal-display module screen for visualization of vocal cords. It is considered an alternative to the flexible fiberoptic endoscope especially in the developing countries where the device cost is the main limiting factor. It has many benefits such as being light weight, easy to clean, durable, chargeable, less expensive and reusable. However newer video stylet devices have not been formally evaluated for tracheal intubation in case of laterally positioned patients.

DETAILED DESCRIPTION:
Following approval from Ethics and Research Committee of Theodor Bilharz Research Institute, the study protocol will be explained to the patients after taking their consent.

Upon arrival to the operating room, a 20 G cannula will be sited intravenously and infusion of Ringer's solution will be started. Intravenous midazolam in a dose of 0.05 mg/ Kg will be given. Then, a five-lead electrocardiogram (GE-Datex Ohmeda 5 lead ECG cable), a pulse oximeter (GE- Datex Ohmeda adult finger spO2 sensor) and a non-invasive blood pressure monitor (GE-Datex Ohmeda NIBP cuff, adult double tube with bag) will be attached to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18- 60 years.
* Both sexes
* American Society of Anesthesiologists(ASA) physical status classes I and II.
* Non-obese patients ( BMI <35)

Exclusion Criteria:

* Difficult intubation; mallampati 3 or 4, Dental abnormalities, Cervical spine pathology that limits neck mobility , obese patients ( BMI ≥ 35) .
* Cardiovascular disease, hypertensive patients, Pregnant and nursing women, High risk of pulmonary aspiration.
* Patients at risk of bleeding either impaired bleeding profile or receiving anticoagulants

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-07-22 (Actual)

PRIMARY OUTCOMES:
Intubation time | up to 1 hour
  (defined as the time when the device is introduced into the mouth till it is removed after the confirmation of correct placement of ETT by the appearance of an optimal waveform on the capnograph

SECONDARY OUTCOMES:
Intubation success rate | up to 1 hour
  Intubation success rate
Number of intubation attempts | up to 1 hour
  Number of intubation attempts
Hemodynamic stability | up to 1 hour
  assessed based on MAP and HR, which will be measured at the following time intervals: before induction of anesthesia at baseline (BA), after induction of anesthesia but before tracheal intubation (T1), and immediately after successful intubation (T2)

CONTACTS AND LOCATIONS:
Overall Officials: Nesrine Elrefai, MD, Principal Investigator — Professor of Anaesthesia, surgical ICU &Pain management; Sohaila Omar, MD, Principal Investigator — Professor of Anaesthesia and surgical ICU; Mohamed Hussien, MD, Study Director — Lecturer of Anaesthesia and surgical ICU
Locations (1):
- Faculty of Medicine, Cairo University., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Still working